CLINICAL TRIAL: NCT02773537
Title: Randomized Comparative Effectiveness Trial of Anesthesia/Analgesia Techniques for Primary Total Knee Arthroplasty
Brief Title: Motor-Sparing Peripheral Nerve Blockade Facilitates Mobility Post Total Knee Arthroplasty: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00042461
Record Dates: First submitted 2016-05-03; First posted 2016-05-16 (Estimated); Results first posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Randomization Group 1 (Active Comparator): Femoral nerve catheter and sciatic nerve block
  Interventions: Drug: Femoral nerve catheter and sciatic nerve block
- Randomization Group 2 (Active Comparator): Adductor canal catheter and selective tibial block
  Interventions: Drug: Adductor canal catheter and selective tibial block
- Randomization Group 3 (Active Comparator): Adductor canal catheter only
  Interventions: Drug: Adductor canal catheter only

INTERVENTIONS:
Drug: Femoral nerve catheter and sciatic nerve block — This nerve block is believed to cause both muscle weakness and numbness. A catheter remains in place for up to 36 hours after surgery for the purpose of adding additional medication should the patient require it. This technique causes both the front and the back of the knee to be numb.
  Arms: Randomization Group 1
Drug: Adductor canal catheter and selective tibial block — This nerve block is believed to cause numbness only, without any muscle weakness. A catheter remains in place for up to 36 hours after surgery for the purpose of adding additional medication should the patient require it to control pain. This technique causes both the front and the back of the knee to be numb.
  Arms: Randomization Group 2
Drug: Adductor canal catheter only — This nerve block is believed to cause numbness only, without any muscle weakness. A catheter remains in place for up to 36 hours after surgery for the purpose of adding additional medication should the patient require it. This technique causes only the front of the knee to be numb
  Arms: Randomization Group 3

SUMMARY:
The primary aim of this pilot study will be to develop a clinically meaningful, patient-centric, and pragmatic protocol to evaluate the comparative effectiveness of different strategies for achievement of the ideal balance between analgesia and functional mobility following total knee arthroplasty (TKA).

DETAILED DESCRIPTION:
Pain management for total knee replacement (TKR) patients has evolved rapidly over the previous decade. The most recent advances in anesthesia include peripheral nerve blockade, which offers the promise of earlier postoperative mobilization in addition to effective pain relief. The rapidity with which these advancements have been adopted seems to have outpaced the science to support them. The result has been the institution of countless combinations of perioperative pain management strategies in centers nationwide with little standardization, consistency, or objective evidence. The extent to which these various strategies achieve safe and effective perioperative pain control or functional preservation remains poorly defined. This prospective randomized control trial will aim to identify meaningful patient-centric outcome measures, differentiate from among three perioperative TKR anesthetic and analgesic strategies, and provide a template for interdisciplinary collaboration among orthopedic surgeons, anesthesiologists, physical therapists, and patients. With the knowledge gained further study will continue to refine the most optimal early pain control protocol.

All primary TKR patients undergoing surgery at the Medical University of South Carolina who are able to receive spinal anesthesia will be randomized prior to surgery to one of three forms of lower limb nerve blockade: 1) Continuous femoral nerve catheter plus single injection sciatic nerve block, 2) Adductor canal catheter plus selective tibial nerve block, 3) Adductor canal catheter alone. All patients will receive additional standardized pain medications as well as early mobilization with physical therapy. The primary outcome measure will be postoperative visual analog pain scale (VAS), with secondary measures to include validated patient-reported outcome measures, objective functional measures (timed-up-and-go (TUG), patient satisfaction scores, length of stay, discharge disposition, and complications. The investigators plan to enroll approximately 90 patients. This will allow us to reach our randomization goal of at least 75 patients while taking into account withdrawals. The 75 patients will be randomized into the three treatment three treatment arms over a 6-month recruitment period, with a 3 month follow-up for patient reported outcome and satisfaction data. A focus group will facilitate patient engagement and provide information for generation of a preference survey to guide future study design.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females 18 years of age or older
* Undergoing elective primary total knee arthroplasty
* Patient is willing and able to give consent and participate

Exclusion Criteria:

* Inability to receive spinal anesthesia or peripheral nerve block
* Non-ambulatory patients
* Non- English speaking patients
* Vulnerable populations including prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Drew, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between October 2015 and August 2016. Patients were approached for participation in the study during their pre-op medical clearance clinic appointment.
Pre-assignment Details: A total of 107 patients undergoing primary TKA met initial eligibility criteria and were offered participation in the trial. 75 total subjects were randomized and considered enrolled to one of three arms of the study. 32 patients were excluded for various reasons prior to randomization.
Groups:
- Femoral Nerve Catheter and Sciatic Nerve Block: Femoral nerve catheter and sciatic nerve block
  Femoral nerve catheter and sciatic nerve block: This nerve block is believed to cause both muscle weakness and numbness. A catheter remains in place for up to 36 hours after surgery for the purpose of adding additional medication should the patient require it. This technique causes both the front and the back of the knee to be numb.
- Adductor Canal Catheter and Selective Tibial Block: Adductor canal catheter and selective tibial block
  Adductor canal catheter and selective tibial block: This nerve block is believed to cause numbness only, without any muscle weakness. A catheter remains in place for up to 36 hours after surgery for the purpose of adding additional medication should the patient require it to control pain. This technique causes both the front and the back of the knee to be numb.
- Adductor Canal Catheter Only: Adductor canal catheter only
  Adductor canal catheter only: This nerve block is believed to cause numbness only, without any muscle weakness. A catheter remains in place for up to 36 hours after surgery for the purpose of adding additional medication should the patient require it. This technique causes only the front of the knee to be numb
Period: Overall Study
Arm/Group | Femoral Nerve Catheter and Sciatic Nerve Block | Adductor Canal Catheter and Selective Tibial Block | Adductor Canal Catheter Only
Started | 25 | 25 | 25
Completed | 25 | 24 | 21
Not Completed | 0 | 1 | 4
Not completed — Lost to Follow-up | 0 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Femoral Nerve Catheter and Sciatic Nerve Block | Adductor Canal Catheter and Selective Tibial Block | Adductor Canal Catheter Only | Total
Number analyzed (Participants) | 25 | 25 | 25 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (6.1) | 65.7 (9.5) | 65.6 (6.8) | 63.8 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 11 | 37
  Male | 10 | 14 | 14 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 9 | 7 | 23
  White | 18 | 16 | 18 | 52
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 25 | 75
Baseline VAS Pain Score [Median (Full Range); unit: Score on a scale] — Pain score on a scale of 0-10 with 0 being the least possible pain and 10 being the worst pain imaginable.
  Score on a scale | 5 [2 to 9] | 6 [0 to 10] | 6 [2 to 10] | 6 [0 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Pain Measurement Via VAS (Visual Analog Scale)
Description: The primary outcome measure will be postoperative visual analog pain scale (VAS) score area under the curve (AUC) for 48 hours, recorded every six hours. Score Scale is 0 (no pain)- 10(most pain). A higher score corresponds to a worse outcome.
Time Frame: 48 hours after procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Femoral Nerve Catheter and Sciatic Nerve Block | Adductor Canal Catheter and Selective Tibial Block | Adductor Canal Catheter Only
Number analyzed (Participants) | 25 | 25 | 25
score on a scale | 4.11 (.43) | 4.68 (.44) | 4.36 (.42)

2. Secondary Outcome: Narcotic Requirements
Description: Narcotic dosages will be measured and reported as oral morphine milligram equivalents.
Time Frame: 48 hours after procedure
Measure: Mean (Inter-Quartile Range); unit: milligrams of morphine equivalents
Arm/Group | Femoral Nerve Catheter and Sciatic Nerve Block | Adductor Canal Catheter and Selective Tibial Block | Adductor Canal Catheter Only
Number analyzed (Participants) | 25 | 25 | 25
milligrams of morphine equivalents | 90 [70 to 125] | 107.5 [84.5 to 142.5] | 107 [77.5 to 162.5]

3. Secondary Outcome: Functional Outcome Measures- Exstension/Knee Buckling
Description: Functional outcome measures will be administered by members of the physical and occupational therapy team, who typically evaluate and treat patients once on the day of surgery and twice daily each day thereafter. They will document the patient's ability to perform independent terminal knee extension and grade knee buckling with ambulation on a scale of 0-2 during each encounter. A grade of 0 indicates no knee buckling, 1 indicates slight buckling, and a grade of 2 represents knee buckling significant enough in the opinion of the physical therapist to require a knee immobilizer while ambulating. I higher score corresponds to a worse outcome. The numbers below in the outcome measure table are the number of patients who achieved terminal knee extension for had ANY knee buckling respectively.
Time Frame: 1-2 days after procedure
Measure: Number; unit: number of participants
Arm/Group | Femoral Nerve Catheter and Sciatic Nerve Block | Adductor Canal Catheter and Selective Tibial Block | Adductor Canal Catheter Only
Number analyzed (Participants) | 25 | 25 | 25
number of participants
  Terminal Knee Extension (Yes) (Post Op. Day 2) | 13 | 15 | 22
  Any Knee Buckling (Yes) (Post Op. Day 1) | 20 | 7 | 8
  Any Knee Buckling (Yes) (PPost Op. Day 2) | 8 | 4 | 1
  Terminal Knee Extension (YES)(Post Op Day 1) | 10 | 16 | 20

4. Secondary Outcome: Functional Outcome Measures- AMPAC (Activity Measure for Post-Acute Care)
Description: Functional outcome measures will be administered by members of the physical and occupational therapy team, who typically evaluate and treat patients once on the day of surgery and twice daily each day thereafter. On the morning of postoperative day #1, the therapist will calculate the Activity Measure for Post-Acute Care (AM-PAC) score. The Activity Measure for Post Acute Care (AM-PAC) measures function in three domains: basic mobility, daily activities,and applied cognitive function. AM-PAC scores in each functional domain have a mean of 50 with a standard deviation of 10 and scores are distributed along a continuum of function. The AM-PAC tracks outcomes as a participant progresses across an episode of care with higher scores indicating an improved level of functioning.
Time Frame: Morning of post-op day 1 - 2 days after procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Femoral Nerve Catheter and Sciatic Nerve Block | Adductor Canal Catheter and Selective Tibial Block | Adductor Canal Catheter Only
Number analyzed (Participants) | 25 | 25 | 25
score on a scale | 15.0 (2.0) | 16.5 (4.0) | 16.0 (2.0)

5. Secondary Outcome: Functional Outcome Measures- TUG (Timed Up and Go)- Distance Walked
Description: Functional outcome measures will be administered by members of the physical and occupational therapy team, who typically evaluate and treat patients once on the day of surgery and twice daily each day thereafter. On the morning of postoperative day #2, the therapist will document distance walked by the patient.
Time Frame: Morning of post-op day 1 - 2 days after procedure
Measure: Mean (Standard Deviation); unit: Feet
Arm/Group | Femoral Nerve Catheter and Sciatic Nerve Block | Adductor Canal Catheter and Selective Tibial Block | Adductor Canal Catheter Only
Number analyzed (Participants) | 25 | 25 | 25
Feet | 80 (102) | 155 (150) | 160 (105)

6. Secondary Outcome: Functional Outcome Measures- TUG (Timed Up and Go)- Time in Seconds
Description: Functional outcome measures will be administered by members of the physical and occupational therapy team, who typically evaluate and treat patients once on the day of surgery and twice daily each day thereafter. On the morning of postoperative day #2, the therapist will document a timed up-and-go test (TUG).
Time Frame: Morning of post-op day 1 - 2 days after procedure
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Femoral Nerve Catheter and Sciatic Nerve Block | Adductor Canal Catheter and Selective Tibial Block | Adductor Canal Catheter Only
Number analyzed (Participants) | 25 | 25 | 25
seconds | 66.1 (32.0) | 61.9 (29.6) | 65.3 (39.3)

7. Secondary Outcome: Patient Reported Pain and Function Outcomes
Description: Short Form Health Survey (SF-12): 12 item abbreviated form of SF-36 survey that provides information about how participants feel, and how well they have been able to perform their usual activities. Transformed physical component summary score (PCS) and transformed mental component summary score (MCS) are derived using the sum of all 12 items and scored onto a 0-100 scale such that a higher score indicates a better health state and better functioning.
  Patient Reported Outcome Measurement Information System (PROMIS): evaluates and monitors physical, mental, and social health. The minimum possible score is 20 and the max is 100.
  Knee injury and Osteoarthritis Outcome Score (KOOS)-Specifically Pain and Symptom Score: A Likert scale is used. All items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale (0=extreme; 100= none).
Time Frame: 6 Weeks after procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Femoral Nerve Catheter and Sciatic Nerve Block | Adductor Canal Catheter and Selective Tibial Block | Adductor Canal Catheter Only
Number analyzed (Participants) | 25 | 25 | 25
score on a scale
  KOOS Pain | 63.3 (19.0) | 57.8 (17.0) | 62.6 (15.8)
  KOOS Symptom | 61.7 (21.8) | 62.6 (16.9) | 58.7 (13.2)
  PROMIS | 37.4 (4.76) | 41.5 (6.35) | 39.2 (6.42)

8. Secondary Outcome: Patient Reported Pain and Function Outcomes
Description: Short Form Health Survey (SF-12): 12 item abbreviated form of SF-36 survey that provides information about how participants feel, and how well they have been able to perform their usual activities. Transformed physical component summary score (PCS) and transformed mental component summary score (MCS) are derived using the sum of all 12 items and scored onto a 0-100 scale such that a higher score indicates a better health state and better functioning.
  Patient Reported Outcome Measurement Information System (PROMIS): evaluates and monitors physical, mental, and social health. The minimum possible score is 20, the maximum is 100.
  Knee injury and Osteoarthritis Outcome Score (KOOS)-Specifically Pain and Symptom Score: A Likert scale is used. All items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale (0=extreme; 100= none).
Time Frame: 3 Months after Procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Femoral Nerve Catheter and Sciatic Nerve Block | Adductor Canal Catheter and Selective Tibial Block | Adductor Canal Catheter Only
Number analyzed (Participants) | 25 | 25 | 25
score on a scale
  KOOS Pain | 66.8 (19.8) | 72.6 (18.4) | 70.5 (17.3)
  KOOS Symptom | 64.3 (19.0) | 71.7 (12.9) | 67.4 (15.8)
  PROMIS | 41.1 (6.92) | 45.4 (7.17) | 44.4 (6.04)

ADVERSE EVENTS:
Time Frame: 3 months post operatively
Arm/Group | Femoral Nerve Catheter and Sciatic Nerve Block | Adductor Canal Catheter and Selective Tibial Block | Adductor Canal Catheter Only
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 2/25 | 5/25 | 2/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Femoral Nerve Catheter and Sciatic Nerve Block (N=25) | Adductor Canal Catheter and Selective Tibial Block (N=25) | Adductor Canal Catheter Only (N=25)
Arthrofibrosis requiring manipulation under anesthesia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flexion Contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Transient thigh muscle spasms, anterior and posterior (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Prolonged wound drainage (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Transient posterior thigh burning (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Persistent decreased sensation, lateral heel Hemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Patellar Tendon rupture after Fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2016-07-13): https://cdn.clinicaltrials.gov/large-docs/37/NCT02773537/Prot_000.pdf